CLINICAL TRIAL: NCT02472392
Title: A Phase I Study to Examine the Toxicity of Allogeneneic Stem Cell Transplantation for Relapsed or Therapy Refractory Ewings
Brief Title: Study To Examine Toxicity Of Allogeneic Stem Cell Transplantation For Relapsed Or Therapy Refractory Ewings Sarcoma
Acronym: Ewing/Allo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.0167
Record Dates: First submitted 2015-06-04; First posted 2015-06-15 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: EWINGS SARCOMA
Keywords: EWINGS, SARCOMA
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Melphalan; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Plan A (Active Comparator): Rabbit anti-thymocyte globulin (ATG) will be given only to unrelated donor transplant recipients at a dose of 3 mg/kg/day I.V. Equine ATG at a dose of 30mg/kg/day may be substituted in the event of severe allergic reaction to the rabbit ATG. Rabbit ATG is only used with recipients of unrelated donor marrow or peripheral blood transplants. Busulfan (BU) will be given at a dose of 0.8 mg/kg IV q 6 hrs. BU doses will be modified based upon pharmacokinetics data to maintain steady state levels of 600-900 ng/dl. Seizure prophylaxis with levetiracetam should begin prior to the 1st dose of BU and stoped 24 hrs after the last dose of BU. Melphalan will be given at a dose of 60 mg/m2 I.V. over 15-20 min per Pediatric SCT Standards of Practice Manual.
  Interventions: Drug: Rabbit anti-thymocyte globulin; Drug: Busulfan; Drug: Melphalan
- Treatment Plan B (Active Comparator): Rabbit anti-thymocyte globulin (ATG) will be given only to unrelated donor transplant recipients at a dose of 3 mg/kg/day I.V. Equine ATG at a dose of 30mg/kg/day may be substituted in the event of severe allergic reaction to the rabbit ATG. Rabbit ATG is only used with recipients of unrelated donor marrow or peripheral blood transplants. Fludarabine will be given at a dose of 30 mg/m2/day IV over 30 mins for 5 doses. Cyclophosphamide will be given at a dose of 50 mg/kg/day IV over 2 hrs for 4 doses.
  Interventions: Drug: Rabbit anti-thymocyte globulin; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rabbit anti-thymocyte globulin — Active treatment
  Other Names: ATG; thymoglobulin
Drug: Busulfan — comparitor
  Other Names: Busulfex; Myleran
  Arms: Treatment Plan A
Drug: Melphalan — comparitor
  Other Names: L-PAM; L-Sarcolysin; Phenylalanine Mustard
  Arms: Treatment Plan A
Drug: Fludarabine — comparitor
  Other Names: Fludara
  Arms: Treatment Plan B
Drug: Cyclophosphamide — comparitor
  Other Names: Cytoxan; Neosar
  Arms: Treatment Plan B

SUMMARY:
The purpose of this study is to examine the toxicity of using allogeneic stem cell transplantation for treatment of subjects with relapsed or refractory ES and rhabdomyosarcoma. This is a nanrandomized two-arm study is designed to determine the safety and incidence of graft versus host disease (GVHD) in patients with relapsed, refractory Ewings sarcoma receiving related and unrelated, allogeneic stem cell transplants.

DETAILED DESCRIPTION:
This study will examine the toxicity of using allogeneic stem cell transplantation for treatment of subjects with relapsed or refractory ES and rhabdomyosarcoma. Donors will consist of either HLA identical or 9/10 (A, B, C, DR, DQ) matched related or unrelated donors. Specifically, we will examine the toxicity of allogeneic stem cell transplant (SCT) in this patient population, as related to incidence of grade 3-4 acute GVHD and the incidence of transplant related mortality at 100 days by using the following treatment plans.

Rabbit anti-thymocyte globulin (ATG; thymoglobulin) will be given only to unrelated donor transplant recipients at a dose of 3 mg/kg/day I.V. for 3 consecutive days (Days -8 to-6). Equine ATG at a dose of 30mg/kg/day may be substituted in the event of severe allergic reaction to the rabbit ATG.

Busulfan (BU) will be given at a dose of 0.8 mg/kg IV q 6 hours, for 16 doses on days -8 through -5. Busulfan doses will be modified based upon pharmacokinetics data to maintain steady state levels of 600-900 ng/dl. Patients should start seizure prophylaxis with levetiracetam prior to the first dose of busulfan and discontinued 24 hours after the last dose of busulfan.

Melphalan will be given at a dose of 60 mg/m2 I.V. over 15-20 min on days -4 through -2 as per Pediatric SCT Standards of Practice Manual.

Fludarabine will be given at a dose of 30 mg/m2/day IV over 30 minutes for 5 doses on days -8 through -4.

Cyclophosphamide will be given at a dose of 50 mg/kg/day IV over 2 hours for 4 doses on days -5 through -2.

Subjects will receive tacrolimus and short course mycophenolate for prohpylactic Therapy incase of Acute Graft-versus-Host Disease.

The following procedures will also be completed throughout this study.

Physical exams and medical histories Frequent blood tests to monitor blood counts, blood chemistries, liver and kidney function Blood tests to determine exposure to various viruses, including viruses that cause hepatitis (inflammation of the liver), the human immunodeficiency virus (HIV, the virus that causes AIDS) and cytomegalovirus Pregnancy test for females of childbearing age Bone Marrow biopsies and aspirates Tests to monitor lung and heart function Evaluations and biopsies to monitor GVHD X-rays, CT or MRI scans for tumor measurements at 1, 3, 6 and 12 months and then at least annually thereafter.

If subjects agree to participate in this research study, they will receive several drugs before the SCT. Various methods will be used to administer medications such asPO, IV, or Central Line placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 0-30 years with relapsed or therapy refractory ES, excluding patients with brain metastases. Patients who have received a prior autologous stem cell transplant are eligible.
2. Related and unrelated marrow and peripheral blood stem donors must be 9/10 or 10/10 (HLA A, B, C, DR, DQ) matched with the recipient

Exclusion Criteria:

1. Organ dysfunction: Patients who have the following levels of organ system dysfunction are not eligible:

   * Cardiac: Ejection Fraction < 50 %
   * Renal: Est. Creatinine Clearance < 50*
   * Hepatic: Bilirubin > 3.0
   * Pulmonary: DLCO < 70 %, or for patient who cannot cooperate with pulmonary function testing, O2 saturation < 95 % on room air.
   * Performance status: Lansky performance < 70; ECOG status > 2 *this is based on the Schwartz formula for children less than 18 years of age, and the Cockcroft - Gault formula, for those > 18 years.[21, 22]
2. Patients with an isolated local recurrence of their tumor (in the site of the primary tumor) > 1 year after completing therapy are excluded, as these patients could be cured with local therapy alone.

3 As a part of the standard of care for pre-transplant evaluation, subjects will be tested for exposure to viral agents such as hepatitis B, C, HTLV-1/2, and HIV. Subjects testing positive for HIV may be rejected as candidates for transplantation, based on the clinical judgment of the stem cell transplant physician

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Toxicity assessed by safety labs and close monitoring from the study staff | Over 5 Years
  This will be assessed by safety labs and close monitoring from the study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lucas, M.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States